CLINICAL TRIAL: NCT07049627
Title: Inflammatory, Nutritional, and Sarcopenia-Based Prediction of Pathological Response in Local Advanced Rectal Cancer: A Regression and AI Approach
Brief Title: AI-Based Prediction of Pathological Response in Rectal Cancer Patients Receiving Total Neoadjuvant Therapy
Acronym: CINR-AI
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, MD, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2024-628
Record Dates: First submitted 2025-06-16; First posted 2025-07-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: Rectal Cancer; Total Neoadjuvant Therapy; Sarcopenia; Artificial Intelligence; Machine Learning
MeSH Terms: conditions — Rectal Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Locally Advanced Rectal Cancer Treated with TNT: This cohort includes 93 patients with clinical stage II-III locally advanced rectal cancer who received total neoadjuvant therapy (TNT), consisting of both systemic chemotherapy and radiotherapy, followed by curative-intent surgery. Patients were retrospectively analyzed to evaluate the predictive role of inflammatory, nutritional, and sarcopenia-based biomarkers on pathological response. No new intervention was administered as part of this study.
  Interventions: Other: Total Neoadjuvant Therapy (TNT)

INTERVENTIONS:
Other: Total Neoadjuvant Therapy (TNT) — Patients included in this retrospective cohort received total neoadjuvant therapy (TNT), consisting of systemic chemotherapy and radiotherapy, followed by curative-intent surgery. No experimental interventions were applied. The analysis focused on evaluating clinical, inflammatory, nutritional, and sarcopenia-based predictors of pathological response.

SUMMARY:
This study aims to better understand how body composition, inflammation, and nutrition affect how rectal cancer responds to treatment. We reviewed data from ninety-three patients who were treated with total neoadjuvant therapy (TNT), which includes both chemotherapy and radiation before surgery. Using blood tests and CT scans, we measured muscle loss (sarcopenia), inflammation, and nutritional status before and after treatment.

This study aims to better understand how body composition, inflammation, and nutrition affect rectal cancer response to treatment. We retrospectively analyzed data from ninety-three patients who received total neoadjuvant therapy (TNT), including both chemotherapy and radiation prior to surgery. Blood tests and CT scans were used to assess inflammation, nutrition, and muscle loss (sarcopenia) before and after treatment. The objective was to identify predictors of complete pathological response. Two novel composite scores were developed from routine lab parameters and tested for their predictive value. Artificial intelligence (AI) was also applied to enhance model accuracy.

This study was conducted at Etlik City Hospital in Ankara, Turkey. No experimental interventions were performed. All data were obtained from routine care, and no additional procedures or patient compensation were involved. The findings may support personalized treatment decisions in rectal cancer.

DETAILED DESCRIPTION:
This is a retrospective observational study that evaluated 93 patients with locally advanced rectal cancer who received total neoadjuvant therapy (TNT) at Etlik City Hospital, Ankara, Turkey, between November 2022 and December 2024. The aim of the study was to investigate whether laboratory markers related to inflammation and nutrition, as well as changes in muscle mass (sarcopenia), could predict treatment response.

Patients who completed at least 12 weeks of chemotherapy and radiotherapy followed by curative surgery were included. Blood samples were used to calculate the C-reactive protein to albumin ratio (CAR) and the systemic immune-inflammation index (SII). Sarcopenia was assessed using contrast-enhanced CT images at the L3 vertebral level, obtained before and after treatment.

Based on these parameters, two composite scores-CINR-pCR and CINR-Ryan-were developed using multivariable logistic regression. The primary outcomes were pathological complete response (pCR) and favorable tumor regression grade (TRG 0-1). Predictive models were constructed using both conventional statistical methods and artificial intelligence (AI)-based algorithms, including Random Forest. Internal validation was performed via cross-validation, and model performance was assessed by area under the curve (AUC), sensitivity, and specificity.

All data used in this study were obtained from existing medical records as part of routine clinical care. No experimental treatments or additional interventions were administered. The results may contribute to optimizing personalized treatment strategies and clinical decision-making in rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* All sexes eligible
* Histologically confirmed clinical stage II-III rectal adenocarcinoma
* Completion of total neoadjuvant therapy (TNT), defined as:
* ≥12 weeks of systemic therapy and
* Radiotherapy (RT) completed
* Curative-intent surgery performed
* Availability of both pre- and post-TNT abdominal CT scans for sarcopenia assessment

Exclusion Criteria:

* Development of distant metastasis during TNT
* Early disease progression
* Missing radiological or pathological data
* Incomplete or non-curative surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective cohort study evaluates pathological response in rectal cancer patients receiving total neoadjuvant therapy (TNT). It integrates systemic inflammation (CAR, SII), nutritional status, and CT-based sarcopenia assessments with both logistic regression and AI (Random Forest) modeling. Two novel composite scores (CINR-pCR and CINR-Ryan) were developed. The study was conducted at Etlik City Hospital, Türkiye, including ninety-three patients between November 2022 and December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | Within 16-24 weeks after TNT completion
  Proportion of patients achieving ypT0N0 following TNT and surgery

SECONDARY OUTCOMES:
Good Pathological Response (TRG 0-1) | Within 16-24 weeks after TNT completion
  Proportion of patients with Tumor Regression Grade 0-1 based on Ryan classification

CONTACTS AND LOCATIONS:
Overall Officials: Galip Can Uyar, MD, Principal Investigator — Ankara Etlik City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik City Hospital, Ankara, Yenimahalle
  - Etlik City Hospital, Ankara, YENİMAHALLE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uyar GC, Basaran BN, Baskurt K, Yesilbas E, Ozkan E, Yucel KB, Altinbas M, Evrimler S, Oksuzoglu OBC, Sutcuoglu O. Predicting Pathologic Response in Locally Advanced Rectal Cancer Using Inflammatory, Nutritional, and Sarcopenia-Based Markers: A Regression and AI-Based Analysis (CINR-AI Study). Clin Colorectal Cancer. 2025 Oct 16:S1533-0028(25)00082-9. doi: 10.1016/j.clcc.2025.10.002. Online ahead of print. PMID 41198426